CLINICAL TRIAL: NCT03999580
Title: A Pragmatic Randomized Controlled Trial on High Dose Vitamin D to Prevent Relapses of Crohn's Disease in Children
Brief Title: The Vitamin D in Pediatric Crohn's Disease ( ViDiPeC-2 )
Acronym: ViDiPeC-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jantchou Prevost (Other)
Responsible Party: Sponsor-Investigator, Jantchou Prevost, Associate Professor of Pediatrics, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-21-2019-2095
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Crohn Disease
Keywords: Crohn; vitamin D; remission; inflammation; tolerance
MeSH Terms: conditions — Crohn Disease; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Time zero for each patient will be the day of randomization. Patients will be randomly assigned (1:1 ratio) in one of two study arms:
  3,000 or 4,000 IU/day, according to the patient body weight, as induction for 4 weeks then 2,000 IU/day as maintenance for 48 weeks. Control: 600 IU/day of Vitamin D as induction (4 weeks) and maintenance (48 weeks).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The vitamin D will be donated by a pharmaceutical company. It will be dispensed in anonymized bottles with the content similar in color and taste in order to keep patients unaware of their allocation. We will implement a number of study maneuvers aimed at minimizing measurement biases. These include: (1) masking of the data; (2) documenting the use of major co-interventions such as other multivitamin supplements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm: (Experimental): Experimental: Vitamin D3 3000 or 4000 UI/day then 2,000 UI/day
  3000 UI or 4,000 UI/day as induction therapy (according to weight) for 4 weeks then 2,000 UI/day as maintenance therapy for 48 weeks.
  The administration of vitamin D will be considered as an adjunct to conventional therapy (corticosteroids, exclusive enteral nutrition or immunosuppressive agents (ISA).
  Interventions: Drug: vitamin D3
- Control Arm: (Active Comparator): Active Comparator: Vitamin D3 600 UI/day then 600 UI/day
  600 UI/day as induction therapy for 4 weeks, then 600 UI/day as maintenance therapy for 48 weeks.
  The administration of vitamin D will be considered as an adjunct to conventional therapy (corticosteroids, exclusive enteral nutrition or immunosuppressive agents (ISA)).
  Interventions: Drug: vitamin D3

INTERVENTIONS:
Drug: vitamin D3 — 3000 or 4000 UI/ day:
  Weight at inclusion < 40 kg : 1 ml per day of the selected concentration at induction and 1ml per day of the selected concentration at maintenance.
  Weight at inclusion ≥ 40 kg : 1 ml per day of the selected concentration at induction and 1 ml per day of the selected concentration at maintenance
  600 UI/ day:
  Weight at inclusion < 40 kg :1 ml per day of the selected concentration (600 IU) at induction and 1 ml per day of the selected concentration (600 IU) at maintenance.
  Weight at inclusion ≥ 40 kg : 1 ml per day of the selected concentration (600 IU) at induction and 1 ml per day of the selected concentration (600 IU) at maintenance
  Other Names: cholecalciferol

SUMMARY:
The purpose of this study is to determine if vitamin D as an adjuvant therapy can improve the outcome (i.e. fewer relapses) and the quality of life, including levels of physical activity, in children diagnosed Crohn's disease (CD).

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory condition affecting all segments of the digestive tract from the mouth to the anus. This condition is associated with an increased risk of relapses throughout the course of the disease. Nearly 25% of patients with Crohn's disease are in the pediatric age range. Many epidemiological data are in favor of an increase incidence of pediatric Crohn's disease. Environmental factors could explain this increased incidence. Among them sunlight exposure and vitamin D deficiency have been suggested by many authors.

Recent studies have described how varying doses of oral vitamin D supplementation can alter serum levels of 25 hydroxyvitamin D (25(OH)D), but no study has specifically addressed the question as to whether vitamin D supplementation can alter the rate of relapse/complications and/or quality of life in children diagnosed with CD.

Current treatments of CD at diagnosis are effective around the time of diagnosis, but in the short and long term, some of these therapies are inefficient or lead to allergic or intolerance reactions. Altogether the rate of relapses in the year after diagnosis is significant. Thus, different therapeutic approaches must be investigated with the aim of lowering the burden of the disease.

From November 2012 to July 2013, we conducted an open label pilot cohort study aiming to investigate the bioavailability and tolerance of high doses of vitamin D3 (3,000 IU or 4,000 IU per day) administered orally as an adjunct therapy in 20 children with newly diagnosed pediatric CD (http://clinicaltrials.gov/ct2/show/NCT01692808). Data from laboratory studies, observational research and pilot trials taken together suggest that vitamin D can be of great importance in the genesis and progression of CD. Vitamin D deficiency could be a true risk factor for disease occurrence and/or relapses. The results of our pilot study demonstrate that in children with active CD at diagnosis, a daily dose of 4,000 IU of vitamin D is well tolerated and quickly increases the blood levels of 25OHD3 to 100 nmol/L or above in 100% of children with CD at diagnosis. Moreover a maintenance dosage of 2,000 IU a day is required (and sufficient) for maintaining this target over several months. Currently there is no adequately powered study in the pediatric CD population exploring the relationship between vitamin D therapy at diagnosis and CD outcomes.

We propose a randomized controlled trial (RCT) to study the efficacy of high-dose oral vitamin D, as adjunct therapy, in children diagnosed CD, to reduce the relapse rate and to improve patients' quality of life.

Primary Efficacy End Point: The proportion of patient with at least one relapse 52 weeks after randomization.

Secondary efficacy endpoint: Quality of life scores, Cumulative steroid dose, Time to first relapse, Duration of corticotherapy, Number of relapses, Number of hospitalizations Safety Endpoint : incidence of hypercalcemia (defined as a corrected serum calcium level >2.65 mmol/L), incidence of hypercalciuria (defined as urinary calcium to creatinine molar ratio ≥1.50), incidence of supra-optimal levels of 25OHD3 as defined by a serum level ≥ 250 nmol/L, rate of study discontinuation due to hypercalcemia or hypercalciuria.

Efficacy Variable: Occurrence of relapse, Time to relapse, Change in QoL score from baseline to 26 weeks, 52 weeks. Change in physical activity score from baseline to 26 weeks, 52 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age at randomization between 4 and 17 years inclusively
2. Pediatric Crohn's Disease Activity Index (PCDAI) ≤ 10 with no clinical symptoms (abdominal pain or blood in the stool) at inclusion
3. Receiving a stable dose for at least 4 weeks of any of the following drugs: Thiopurines, Methotrexate, or TNF-α inhibitors (Infliximab/Adalimumab)
4. Dosage of fecal calprotectin lower than 250 µg/g stool at inclusion.

Exclusion Criteria:

1. History of surgery resulting in a permanent colostomy or ileostomy (because of the inability to calculate PCDAI at baseline)
2. Patients who have already been included in the pilots vitamin D trials
3. Patients actively enrolled in other CD drug trials.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 316 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Relapse | Within 52 weeks after randomization in the study
  A relapse is defined as the occurrence of clinical symptoms (> 2 bowel movements per day, abdominal pain, fever, weight loss, perianal disease or extra-intestinal symptoms) and a pediatric Crohn's disease Activity Index (PCDAI) less than 10.
  The PCDAI is a validated and reproducible tool that was developed by consensus at a meeting of pediatric (Inflammatory bowel disease) IBD experts and subsequently validated in 12 North American institutions. It includes 11 domains, with clinical symptoms, physical examination, laboratory parameters, and growth.
  The PCDAI score can range from 0-100, with higher scores signifying more active disease. A score < 10 is consistent with inactive disease; 11-30 indicates mild disease; > 30 suggests moderate to severe disease. The PCDAI has been used in many pediatric trials.

SECONDARY OUTCOMES:
Lapse of time from randomization to first relapse | From date of randomization until the date of first relapse, assessed up to 52 weeks after randomization in the study
  numbers of days between the randomisation and the first relapse
Number of relapses per patient per year | Within 52 weeks after randomization in the study
  numbers of relapses during the entire study
Number of hospitalizations per year | Between randomization and Week 52
  numbers of hospitalizations during the entire study
Improvement of the Quality of life | At week 26 and week 52
  As measured by the IMPACT III questionnaire. IMPACT III is a validated questionnaire that assesses disease-related quality-of-life in multiple domains of care in pediatric IBD (bowel symptoms; systemic symptoms; emotional functioning; functional/social impairment; body image; test-treatments). Overall scores for IMPACT III range from 35 to 175 with higher scores associated with better quality of life

OTHER OUTCOMES:
Change in the level of physical activities | Between randomization and 52 weeks
  As measured by the Canadian Health Measures Survey - Children's Physical Activity. It includes 35 short questions. This is a questionnaire that has already been used by Canadian children. The responses will be converted into metabolic equivalents of tasks (METS) by using validated tables. Any activity ≥ 3 METS will be classified as moderate-to-vigorous physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Prevost Jantchou, MD,PhD, Principal Investigator — St. Justine's Hospital
Locations (7):
- Canada (7):
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jantchou, P., Mailhot, G., Ezri, J., Le Deist, F., Deslandres, C., & Delvin, E. (2014). P-102: Bioavailability and tolerance of high doses vitamin D in children with newly diagnosed Crohn's disease. Journal of Crohn's and Colitis, 8, S432. doi:10.1016/s1873-9946(14)50130-4
- [Background] Jantchou P, Clavel-Chapelon F, Racine A, Kvaskoff M, Carbonnel F, Boutron-Ruault MC. High residential sun exposure is associated with a low risk of incident Crohn's disease in the prospective E3N cohort. Inflamm Bowel Dis. 2014 Jan;20(1):75-81. doi: 10.1097/01.MIB.0000436275.12131.4f. PMID 24247650